CLINICAL TRIAL: NCT05279222
Title: The Influence of Surgical Correction of Foot Deformity on the Effect of Gait Training on Gait Capacity in Chronic Stroke Patients
Brief Title: Window of Trainability in Relation to Surgical Correction of Foot Deformity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled in the study within an inclusion period of 8 months
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 993_Pes_equinovarus_training
Record Dates: First submitted 2022-02-04; First posted 2022-03-15 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- gait training (Experimental)
  Interventions: Other: Gait adaptability training

INTERVENTIONS:
Other: Gait adaptability training — All patients will receive two gait training interventions, each consisting of twelve one hour training sessions. The training sessions will be focussed on improving gait capacity.

SUMMARY:
Background: Stroke is the leading cause of disability in the western world. In chronic stroke patients, foot deformity such as pes equinovarus is among the most important underlying motor deficits, due to imbalance of muscle strength and activity around the ankle and tarsal joints. Both nationally and internationally, there is relative underuse of surgical treatment options, although in our clinical experience this often has the best outcome. In addition to positive clinical experiences with surgical interventions, we have experienced that before surgery, there is limited effect of gait training on gait capacity. However, we have experienced that after surgery, the restored normal ankle-foot position creates a new window for training opportunities to further improve gait capacity. Therefore, in this exploratory proof of principle study we aim to investigate the effect of surgical correction of post-stroke foot deformity on the (potential) improvement of gait capacity after gait training. Based on clinical experiences, we expect that after surgery, gait training results in a larger improvement in gait capacity compared to before the surgical intervention due to the increased possibilities to improve balance control.

Objective: The primary objective of this study is to compare the effect of gait training on gait capacity (stepping performance, gait adaptability and dynamic balance) before and after surgical correction of post-stroke foot deformity.

Study design: Exploratory proof of principle study with repeated-measures. Study population: Fifteen stroke patients with disabling foot deformity will be recruited from the Gait Expertise Center (LEC) of the Sint Maartenskliniek and Radboudumc.

Intervention: All patients will receive two gait training interventions, each consisting of twelve one hour training sessions. The training sessions will be focussed on improving gait capacity.

Main study parameters/endpoints: Primary outcomes will be gait adaptability as measured with the Emory Function Ambulation Profile (E-FAP), stepping performance as measured with the Timed-Up-And-Go test (TUG) and dynamic balance as measured with the Margin of Stability (MoS).

ELIGIBILITY:
Inclusion Criteria:

* > 6 months post onset
* 18 years or older
* Functional Ambulation Classification (FAC) => 3: the patient is able to walk without physical support
* Will undergo a surgical correction of foot deformity

Exclusion Criteria:

* suffers from any other disorder that seriously affects gait capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Emory Functional Ambulation Profile score | 20 minutes
  Measure for gait adaptability. The E-FAP consists of five subtasks: a 5-meter walk test on a hard-surfaced floor, a 5-meter walk test on a carpeted floor, an up and go task, an obstacle course, and ascent and descent of four stairs. The subtasks will be completed according to the sequence above and the time it takes to complete each subtask will be recorded. A standardized E-FAP protocol will be used to assess the subtasks of the E-FAP.
Margin of Stability (MoS) (cm) | 30 minutes
  Measure for gait capacity. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.
Timed-Up-And-Go test (TUG) score (s) | 1 minute
  Measure for gait capacity.

SECONDARY OUTCOMES:
Walking Adaptability Ladder Test score | 5 minutes
  Measure for gait adaptability. For this test, a standardized ladder is placed on the floor. It consists of 17 rectangular stepping targets that gradually decrease 2 cm in length (range 64-32 cm). Participants start stepping in the largest target and walk as fast as possible to the other side, turn and hit the targets in reverse order while avoiding the ladder rungs. The instructions are to perform the test as fast as possible, without making foot placement errors. The test is timed: a faster time is indicative of a better gait adaptability. Participants perform the test four times, first twice with one foot per target and, thereafter, twice with both feet in one target. A time penalty of 0.5 s is added each time a participant makes a foot placement mistake.
Modified Dynamic Gait Index score | 20 minutes
  Measure for gait adaptability. The modified Dynamic Gait Index consists of 8 subtasks: usual pace, change pace, horizontal head turns, vertical head turns, pivot turn, stepping over obstacles, stepping around obstacles and stairs. The subtasks will be performed according to the mDIG protocol. The time to complete each subtask will be recorded and used as outcome measure.
Lyapunov exponent (-) | 30 minutes
  Measure for dynamic balance. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.
Foot placement estimator (cm) | 30 minutes
  Measure for dynamic balance. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.
Distance between extrapolated center of mass (XCoM) and center of pressure (CoP) in anterior-posterior (AP) and medio-lateral (ML) direction (cm) | 30 minutes
  Measure for dynamic balance. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.
Center of mass (CoM) - center of pressure (CoP) inclination angles (degrees) | 30 minutes
  Measure for dynamic balance. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.
Step width variability (cm) | 30 minutes
  Measure for dynamic balance. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.
Step time variability (s) | 30 minutes
  Measure for dynamic balance. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.
Activities-specific Balance Confidence Scale (ABC Scale) | 10 minutes
  Measure for dynamic balance.
Walking speed (m/s) | 30 minutes
  Measure for gait capacity. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.
Hip-knee-ankle-foot kinematics (degrees) | 30 minutes
  Measure for gait capacity. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.
Peak ankle moment (Nm) | 30 minutes
  Measure for gait capacity. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.
Peak ankle power (W) | 30 minutes
  Measure for gait capacity. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.
Mini-BESTest score | 20 minutes
  Measure for gait capacity.
Activity during the training sessions (minutes) | 1 minute
  Measured by the Polar A360 activity tracker.
Logbook training sessions (training excercises) | 15 minutes
  In the logbook, the therapist describes the exact tasks that are performed during the training sessions.
Step length (m) | 30 minutes
  Measure for gait capacity. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.
Cadence (steps/minute) | 30 minutes
  Measure for gait capacity. Measured by using the Gait Real Time Analysis Interactive Lab as a measurement device.

OTHER OUTCOMES:
Sex (man/ woman) | 0 minutes
Age (years) | 0 minutes
Height (cm) | 1 minute
Weight (kg) | 1 minute
Body Mass Index (BMI) | 0 minutes
  Calculated with the weight and height

CONTACTS AND LOCATIONS:
Locations (1):
- Netherlands, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided